CLINICAL TRIAL: NCT03625583
Title: A Multi-centre Study of Epidemiology, Characteristics, Treatment and Outcome of Chronic Myeloid Leukaemia in Adults in Hong Kong
Brief Title: The Hong Kong CML Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Yok-lam Kwong, Chair Professor, The University of Hong Kong
Other Study IDs: QMH-CML-003
Record Dates: First submitted 2018-07-25; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic myeloid leukaemia: chronic myeloid leukaemia diagnosed from 2007 - 2017

SUMMARY:
Chronic myeloid leukaemia (CML) is a malignant disorder of the haematopoietic system. It is characterized by the chromosomal translocation between chromosomes 9 and 22, resulting in the formation of the Philadelphia chromosome which contains the BCRABL1 fusion gene. The projected prevalence of CML is rising steadily, due to the significantly improved survival of CML patients and that the incidence rate increases with age. The efficacious yet costly tyrosine kinase inhibitors pose a significant financial burden to both patients and the health care system, while they carry their own side effects and long-term risks. This study aims to set up a local disease registry of CML to improve the knowledge concerning this disease, including epidemiology,characteristics and treatment outcome of CML in Hong Kong,as well as long-term safety and toxicities of therapeutic agents.

DETAILED DESCRIPTION:
Chronic myeloid leukaemia (CML) is a malignant disorder of the haematopoietic system characterized by the presence of the Philadelphia chromosome arising from t(9;22)(q34;q 11).The annual incidence of CML is reported to be around 1-2 cases per 100,000 population.In Hong Kong, the age-standardised incidence rate of CML has remained static in recent years.

However, as the incidence of CML increases with age and Hong Kong has an ageing population, the crude incidence rate is expected to follow a rising trend. On the other hand, the prognosis of CML patients has improved significantly since the advent of tyrosine kinase inhibitors (TKis) more than two decades ago. With the efficacious TKis, CML has changed from a deadly cancer to a treatable chronic condition. It has been shown that life expectancy of CML patients is approaching that of the general population now.The prevalence of CML is expected to rise considerably in view of the increasing incidence in an ageing population and improved prognosis. The Hong Kong Cancer Registry only provides data on the incidence rates of cancers but it has yet to provide cancer prevalence data. A clinical registry is "an organized system that uses observational study methods to collect uniform data to evaluate specific outcomes". A disease registry specifically designed for CML would provide more accurate and comprehensive data and allow an in-depth study of the epidemiology and characteristics of CML in Hong Kong.

At present,there are three TKis approved for front-line treatment of newly diagnosed chronic-phase CML,viz.,imatinib, nilotinib and dasatinib.lmatinib is a first-generation TKI while nilotinib and dasatinib are second-generation TKis (2G-TKI) . Nilotinib and dasatinib demonstrate better in vitro efficacy and achieve molecular responses faster and deeper than imatinib,but these drugs not been proven superior to imatinib in conventional clinical endpoints including overall survival and progression-free survival.Besides, nilotinib and dasatinib are not without side effects and their long-term safety profiles are unclear. For example, nilotinib is associated with increased cardiovascular risk while dasatinib often leads to pleural effusion and less frequently,pulmonary hypertension.The safety of imatinib has been well established over the past 15 years and its side effects are generally considered tolerable. However, the generic formulation of imatinib has been recently introduced to public hospitals and substituted for branded imatinib in CML patients. There have been reports that patient switching to generic imatinib develop adverse drug reactions not experienced with branded imatinib. Other less commonly used therapeutic agents include bosutinib and ponatinib, which still play an important role in the management of CML. Therefore, it is important to determine the "real-world" clinical effectiveness of various drugs, and monitor their side effects and long-term toxicities in a population-based approach.

As physicians in Hong Kong are facing a growing patient population on long-term TKI,the demand on health care services and financial burden of drug costs will escalate accordingly. lt is pivotal for the investigators to understand the disease and patients in the locality better by systematic data collection, in order to improve quality of care, allow service planning and facilitate medical research and advances .

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or above
2. Diagnosed with Philadelphia chromosome positive and/or BCR-ABLl positive chronic myeloid leukaemia in all phases
3. Managed in any of the participating centres in the period of 2007 to 2017

Exclusion Criteria:

1) Patients less than 18years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Descriptive statistics will be used to analyse the characteristics of the CML cohort. Categorical data will be presented with frequency, percentage and 95% confidence interval. Quantitative variables will be presented with median and range, mean and standard deviation when relevant. Survival data will be analysed by the Kaplan-Meier method and competing risks methods. A P value of less than 0.05 will be considered statistically significant. All analyses will be performed using SPSS version 24 and Rsoftware version3.3.2.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Demographics | January 2007 to December 2017
  percentage of ethnic distribution
Age | January 2007 to December 2017
  percentage of age distribution
Etiology | January 2007 to December 2017
  percentage of etiology
Clinical features | January 2007 to December 2017
  percentage of clinical features
Sex | January 2007 to December 2017
  ratio of male to female patient

SECONDARY OUTCOMES:
number of CML patients in Hong Kong | up to 10 years
  Estimated prevalence of CML in Hong Kong
number of newly diagnosis CML patient each year | up to 10 years
  Estimated incidence of CML in Hong Kong
Current treatment pattern of CML | up to 10 years
  Current treatment pattern of CML
record AE of each treatment | up to 10 years
  Safety data ofTKI
disease free and survival free | up to 10 years
  Treatment outcome of CML patients
disease free and survival free data in advanced phases (accelerated and blast phases) | up to 10 years
  Outcome of patients in advanced phases (accelerated and blast phases)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Carol Cheung, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided